CLINICAL TRIAL: NCT01368068
Title: Double-Blind Randomised Investigation of Tibolone or Escitalopram in First Onset Perimenopausal Depression
Brief Title: Investigation of Tibolone and Escitalopram in Perimenopausal Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Professor, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 161/11
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Perimenopausal Depression
Keywords: Perimenopause; Depression
MeSH Terms: conditions — Depression | interventions — tibolone; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tibolone (Experimental): Subjects will take 2.5mg of oral Tibolone daily for the duration of the 12 week trial.
  Interventions: Drug: Tibolone
- Escitalopram (Active Comparator): 10mg of escitalopram will be taken by participants daily for the duration of the 12 week trial period.
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Placebo arm containing sweetener has been approved and will be used as placebo arm.
  Interventions: Drug: Natvia

INTERVENTIONS:
Drug: Tibolone — 2.5mg/oral/daily
  Other Names: Livial
  Arms: Tibolone
Drug: Escitalopram — 10mg/oral/daily
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Natvia — serving size: 0.09g per tablet
  Other Names: Natvia Natural Sweetener
  Arms: Placebo

SUMMARY:
Many perimenopausal women experience severe mood symptoms for the first time in their life, with no past psychiatric history. The importance of clearly identifying and treating a disorder that is increasingly referred to as "perimenopausal depression" is highlighted by the wide-reaching impact this can have on the lives of women suffering from it. This is not a minor or short term mood disturbance; it is a severe depressive illness, needing effective and early treatment. Relationships, employment, participation in social roles and individual well-being can all be disrupted by the combination of the mood, hormonal and physical changes associated with the transition to menopause. The term "perimenopausal depression" denotes the onset of depression coinciding with the onset of reproductive hormone changes.

Many women with this type of depression experience serious and long term debilitating symptoms. Treatment commonly draws on traditional approaches for the management of major depression including the use of antidepressants such as selective serotonin reuptake inhibitors (SSRIs) as the first line response. However, standard treatment of perimenopausal depression using antidepressants has only shown small improvements at best and at worst, is associated with severe side effects. Some SSRIs have been shown to be less effective in postmenopausal women compared to child bearing age women. Hormone treatments directly targeting the fluctuating reproductive hormone systems (in particular estrogen) through the administration of compounds such as tibolone, have significant potential as a better overall treatment.

To date, there is still a lack of clear clinical evidence about the best approach for the biological treatment of women with perimenopausal depression. The project we now propose to conduct is a 12-week randomised controlled trial (RCT) of 2.5 mg/day tibolone compared to 10mg/day of escitalopram (an SSRI that has targeted serotonin action)compared to placebo to discover the best treatment approach for a hitherto understudied depression that affects a large proportion of women in their late forties and fifties.

DETAILED DESCRIPTION:
All women experience menopause and a significant number suffer from ongoing, severe depression beginning with the major hormone fluctuations in this middle stage of life. The number of women experiencing menopause related major depression and the impact of this depression on the woman's life, work and her family are grossly underestimated. We propose to conduct a clinical trial of a new hormone treatment for women with severe depression related to menopause, compared with standard antidepressant medication.

Longitudinal epidemiological studies have shown that many women experience significant physical and psychological changes as they approach menopause and for a long time following. Vasomotor symptoms (such as hot flushes, night sweats), sleep disturbances and changes in libido are common, and impact significantly on the quality of life, social and personal well-being. However, the major reason that many women seek help from menopause clinics or their doctors, is for depression and anxiety symptoms.

Many perimenopausal women experience severe mood symptoms for the first time in their life, with no past psychiatric history. The importance of clearly identifying and treating a disorder that is increasingly referred to as "perimenopausal depression" is highlighted by the wide-reaching impact this can have on the lives of women suffering from it. This is not a minor or short term mood disturbance; it is a severe depressive illness, needing effective and early treatment. Relationships, employment, participation in social roles and individual well-being can all be disrupted by the combination of the mood, hormonal and physical changes associated with the transition to menopause. The term "perimenopausal depression" denotes the onset of depression coinciding with the onset of reproductive hormone changes.

Many women with this type of depression experience serious and long term debilitating symptoms. Treatment commonly draws on traditional approaches for the management of major depression including the use of antidepressants such as selective serotonin reuptake inhibitors (SSRIs) as the first line response. However, standard treatment of perimenopausal depression using antidepressants has only shown small improvements at best and at worst, is associated with severe side effects. Some SSRIs have been shown to be less effective in postmenopausal women compared to child bearing age women. Hormone treatments directly targeting the fluctuating reproductive hormone systems (in particular estrogen) through the administration of compounds such as tibolone, have significant potential as a better overall treatment.

To date, there is still a lack of clear clinical evidence about the best approach for the biological treatment of women with perimenopausal depression. The project we now propose to conduct is a 12-week randomised controlled trial (RCT) of 2.5 mg/day tibolone compared to 10mg/day of escitalopram (an SSRI that has targeted serotonin action) compared to placebo to discover the best treatment approach for a hitherto understudied depression that affects a large proportion of women in their late forties and fifties.

ELIGIBILITY:
Inclusion Criteria:

* Females who are currently physically well and between 45 and 55 years of age
* Current DSM-IV diagnosis of depression disorder
* Able to give informed consent
* Perimenopausal as determined by symptom profile on the Stages of Reproductive Aging Workshop and gonadal hormonal profile

Exclusion Criteria:

* Known abnormalities in the hypothalamic-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, active or past history of a venous thromboembolic event, breast pathology, undiagnosed vaginal bleeding or abnormal Pap smear results in the previous 2 years.
* Patients with any significant unstable medical illness such as epilepsy and diabetes or known active cardiac, renal or liver disease; or the presence of illness causing immobilisation.
* Patients receiving treatment for depression including antidepressant medications, electroconvulsive therapy (ECT) / Transcranial Magnetic Stimulation (TMS), formal psychotherapy or counselling, within the past 6 months
* Patients experiencing severe melancholia, neurovegetative symptoms or current suicidality necessitating acute hospitalisation or intensive psychiatric treatment.
* Patients with psychotic symptoms or past history of severe mental illness including schizophrenia, and bipolar disorder.
* Use of any form of estrogen, progestin or androgen as hormonal therapy, or antiandrogen including tibolone or use of phytoestrogen supplements as powder or tablet
* Pregnancy / Lactation
* Smoking cigarettes and other nicotine products.
* illicit drug use and more than 3 standard drinks per day

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale | Baseline, then at weeks 2, 4, 8 and 12.
  A 10-item clinician rated scale validated to be most strongly sensitive to change in depression associated with treatment. This scale will be used to measure change in depression associated with treatment at weeks 2, 4, 8 and 12 compared to baseline.

SECONDARY OUTCOMES:
Short Form-36 Health Survey (SF-36) | Baseline and 12
  A 36 item self report measure that assesses: physical health and bodily pain; vitality, social functioning; role limitations due to emotional problems; and mental health. This scale will be used to assess the changes to various domains of self-reported health from baseline compared to visits at baseline and week 12.
Pittsburgh Sleep Quality Index | Baseline and 12.
  A valid and reliable 19-item self report index measuring sleep quality, latency, duration, disturbances, and daytime dysfunction. This scale will be used to measure different domains of sleep quality at visits occurring at week baseline and week 12 compared to initial baseline measurement.
Adverse Symptoms Checklist | Weeks 2, 4, 8 and 12
  A 22 item checklist of general adverse symptoms experienced. This scale will be used to measure adverse symptoms experienced by participants at weeks 2, 4, 8 and 12 compared to baseline.
Beck Depression Inventory Scale | Baseline and week 12
  A subjective rating scale that compliments the MADRS and will be used at baseline and week 12 visits throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, PhD,FRANZP, Principal Investigator — Monash Alfred Psychiatry Research Centre
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia